CLINICAL TRIAL: NCT06641648
Title: A Phase I Single-arm Clinical Study of Donor NK Cells Infusion Combined with Low-dose Interleukin-2 in the Treatment of Acute Myeloid Leukemia Relapse After Allogeneic Hematopoietic Stem Cell Transplantation.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yujun DONG, chief of department of hematology, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUFH JDCO2
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia (AML) Relapse; NK Cell
Keywords: AML; relapse; allogeneic hematopoietic stem cell transplantation.; NK cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NK cell treatment in AML replase after HSCT (Experimental): The relapsed AML patients will receive donor NK cells injections for a total dose of twice per 2 weeks up to 3 dose levels (1.0×108 cells/dose，5.0×108 cells/dose，2.0×109 cells/dose), followed by low-dose interleukin-2 (1mIU ih, Qd) for 28 days.
  Interventions: Drug: NK cell

INTERVENTIONS:
Drug: NK cell — Drug: Donor NK cells injection is a non-genetically modified natural killer cells therapy derived from a healthy donor.

SUMMARY:
This is a single-centre, single-arm, open-label, early clinical study to evaluate the safety, tolerability and preliminary efficacy of donor NK cells injection combined with low-dose interleukin-2 in the treatment of acute myeloid leukemia (AML) relapse after allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
This is a dose-escalation study of non-genetically modified natural killer cells derived from a healthy donor. The relapsed AML patients after allo-HSCT will receive donor NK cells injection s followed by low-dose interleukin-2. No graft-versus-host disease (GVHD) prevention will be conducted before or after infusion. Dose-limiting toxicity, incidence of adverse events, disease response and PK/PD will be detected post-infusion.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 18 years old, no gender or race; 2.Expected survival period ≥ 3 months; 3.Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2; 4.The diagnosis of AML who received allo-HSCT, and met the following criteria: A. Diagnostic criteria for relapsed AML: after complete remission (CR), leukemia cells reappeared in peripheral blood or blast cells in bone marrow ≥ 5% (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia cell infiltration; B. Minimal Residual Disease (MRD) positive only or relapse: Patient is minimal residual disease (MRD) positive, as assessed on bone marrow aspirate (BMA) by Multiparameter Flow Cytometry (MFC) at time of Treatment Eligibility assessment; C. Degree II and above acute graft-versus-host disease did not occur after transplantation; D. Available allogeneic hematopoietic stem cell transplant donors. 5. Adequate organ function: A. Liver function: ALT≤3×ULN, AST≤3×ULN, total bilirubin≤2×ULN; B. Coagulation function: international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤ 1.5×ULN; C. Renal function: serum creatinine≤1.5×ULN or creatinine clearance rate ≥30mL/min; D. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 45%; 6. Women of child-bearing potential and all male participants must use effective methods of contraception for at least 12 months after infusion.; 7. Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* 1. Central nervous system involved; 2. Patients who received the following anti-tumor therapies prior to infusion: A. Systemic use of hormones within 3 days prior to infusion (except for patients with inhaled corticosteroids); B. Systemic anti-tumor therapy within 2 weeks or within 5 drug half-lives (whichever is shorter); C. Radiotherapy within 4 weeks; D. DLI within 6 weeks; E. Intrathecal injection within 1 week; F. Received CAR-T, CAR-NK or other modified cell therapy within 6 months; 3. Any active infection requiring systemic therapy by intravenous infusion within 14 days prior to the first dose of study drug, including: HBV, HCV, HIV, syphilis infection, or active pulmonary tuberculosis.

  4. History of hypersensitivity reactions to murine protein-containing products, or macromolecular biopharmaceuticals such as antibodies or cytokines; 5. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 years after enrollment; 6. Women who are pregnant (urine/blood pregnancy test positive) or lactating; 7. Suffering from a serious autoimmune disease or immunodeficiency disease; 8. Known alcohol dependence or drug dependence; 9. According to the investigator's judgment, the patient has other unsuitable grouping conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 1 month
  Dose limiting toxicities (DLTs)
Treatment-related adverse events | 1 month
  Treatment-related adverse events

SECONDARY OUTCOMES:
Complete response (CR) | 3 months
  Complete response (CR)
Proportion of subjects with minimal-residual disease (MRD) negative response | 3 months
Peak levels of donor NK cells (maximum concentration or Cmax) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yujun Dong, Docter, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No